CLINICAL TRIAL: NCT03587181
Title: Investigation of Substrates Associated With the Recurrence of Atrial Fibrillation After PV Cryoablation
Acronym: SubstrateAF
Status: Completed | Type: Observational
Sponsor: National Research Center for Preventive Medicine (Other Government)
Collaborators: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Sponsor
Organization: National Medical Research Center for Therapy and Preventive Medicine (Other Government)
Other Study IDs: 01-04/18
Record Dates: First submitted 2018-07-02; First posted 2018-07-16 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Atrial Fibrillation
Keywords: Cryoballoon, Cryoablation, biobanking, Loop recorder, biopsy
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Before intervention blood samples will be collected for biobank storage. It is planned to assess levels of NT-proBNP, high-sensitive CRP, TNF, IL1B, FABP, MMP1, MMP3, MMP9, TGF-beta1, TIMP-1, FGF-9.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Cryoablation of the pulmonary veins and myocardial biopsy — Before intervention blood samples will be collected for biobank storage. After left atrial appendage thrombus exclusion, a cardiac biopsy from intraventricular and interatrial septum will be performed. PV isolation will be performed with cryoablation. Successful PV isolation will be confirmed by the confirmation of bi-directional block. Phrenic nerve function will be assessed in a standard fashion during intervention of the right PVs using high output phrenic nerve pacing from the superior vena cava. Loop recorder implantation will be performed during the same procedure.
  In patients with recurrent atrial tachyarrhythmias an EP study will be performed to assess the mechanism of recurrence. PV reconnections will be re-isolated and linear lesions performed as required.
  Other Names: loop recorder implantation

SUMMARY:
The two main mechanisms for atrial fibrillation (AF) recurrence after cryoablation include Pulmonary vein (PV) reconnection and the presence of non-PV associated arrhythmic focuses. The aim of this study is to investigate the prevalence of each mechanism and if biomarkers may be used to predict of these events.

Eighty patients with paroxysmal or persistent AF will undergo PV isolation with cryoablation followed by loop recorder implantation. Patients in whom atrial tachyarrhythmias recur during 12 months follow-up (outside of the 3-month post procedure blanking window) will be offered a second electrophysiology study (EP) study to assess PV isolation and non-PV focuses and further ablation performed as required.

At baseline blood samples will be taken to investigate the correlation between specific biomarkers and both the incidence and type of recurrence. The correlation between recurrence of atrial tachyarrhythmias due to non-PV associated arrhythmic focuses and elevated baseline levels of NT-ProBNP, CRP, TNF, MMP1 will be pre-specified.

40 consecutive patients will have a biopsy taken from the intraventricular and interatrial septum to investigate the correlation between myocardial inflammation, the presence of fibrosis and recurrence of atrial tachyarrhythmias. Correlation between biomarkers of inflammation and biopsy-proven myocardial inflammation or fibrosis will be assessed.

DETAILED DESCRIPTION:
The two main mechanisms for atrial fibrillation (AF) recurrence after cryoablation include Pulmonary vein (PV) reconnection and the presence of non-PV associated arrhythmic focuses. The aim of this study is to investigate the prevalence of each mechanism and if biomarkers may be used to predict these events.

Eighty patients with paroxysmal or persistent AF will undergo PV isolation with cryoablation followed by loop recorder implantation. Patients in whom atrial tachyarrhythmias recur during 12 months follow-up (outside of the 3-month post procedure blanking window) will be offered a second EP study to assess PV isolation and non-PV focuses and further ablation performed as required. Recurrence will be defined as an episode of atrial tachyarrhythmia (AF, atypical atrial flutter, or atrial tachycardia) on loop recorder with a duration greater than 30 seconds or ECG document atrial tachyarrhythmia. The incidence of atrial tachyarrhythmia recurrence, and its association with symptoms after the index PV cryoballoon isolation, will be assessed.

At baseline blood samples will be taken to assess levels of N-terminal pro brain natriuretic peptide (NT-proBNP), High-sensitivity C-reactive protein (high-sensitive CRP), Tumor Necrosis Factor (TNF), Interleukin 1 beta (IL1B), Fatty acid binding protein (FABP), Matrix metalloproteinase-1 (MMP1), Matrix metalloproteinase-3 (MMP3), Matrix metalloproteinase-9 (MMP9), Transforming growth factor beta 1 (TGF-beta1), Tissue inhibitor of metalloproteinases 1 (TIMP-1), Fibroblast growth factor 9 (FGF-9). Correlation between recurrence of atrial tachyarrhythmias due to non-PV associated arrhythmic focuses and elevated baseline levels of NT-ProBNP, CRP, TNF, MMP1 will be pre-specified. We will look with receiver operating characteristic (ROC) curve analysis the level of biomarkers which predict recurrence of atrial tachyarrhythmias with the best ratio between sensitivity and specificity.

40 consecutive patients will have a biopsy taken from the intraventricular and interatrial septum to investigate the correlation between myocardial inflammation, the presence of fibrosis and recurrence of atrial tachyarrhythmias. Correlation between biomarkers of inflammation and biopsy-proven myocardial inflammation or fibrosis will be assessed.

ELIGIBILITY:
Inclusion Criteria:

• Patient with paroxysmal/persistent atrial fibrillation (EHRA scale 2b-4)

Exclusion Criteria:

* prior interventions for AF
* permanent AF
* contraindications to oral anticoagulation or heparin
* chronic kidney disease requiring dialysis
* untreated hypo- or hyperthyroidism
* breast feeding
* pregnancy
* chronic kidney disease requiring dialysis
* decompensated heart failure
* stroke within the last 3 months
* myocardial infarction within the last 3 months
* Percutaneous coronary intervention or Coronary Artery Bypass Grafting within the last 3 months
* active myocarditis
* artificial valve replacement surgery
* severe mitral or aortic stenosis
* coronary artery disease requiring revascularization
* heart transplant

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 18-80 years old with symptomatic paroxismal or persistant atrial fibrillation (EHRA scale 2b-4)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-04-03 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
Atrial tachyarrhythmia recurrence | 1 year
  Atrial tachyarrhythmias recurrence by ECG, Holter monitoring or loop recorder after 3 months of blanking period

SECONDARY OUTCOMES:
The prevalence of PV reconnection and non-PV focuses as substrate of atrial tachyarrhythmia after cryoablation | 1 year
The difference in baseline NT-ProBNP levels between those patients with recurrence of atrial tachyarrhythmias due to non-PV associated arrhythmic focuses and those without at 12 months | 1 year
The difference in baseline CRP levels between those patients with recurrence of atrial tachyarrhythmias due to non-PV associated arrhythmic focuses and those without at 12 months | 1 year
The difference in baseline TNF levels between those patients with recurrence of atrial tachyarrhythmias due to non-PV associated arrhythmic focuses and those without at 12 months | 1 year
The difference in baseline MMP1 levels between those patients with recurrence of atrial tachyarrhythmias due to non-PV associated arrhythmic focuses and those without at 12 months | 1 year
The difference in baseline NT-ProBNP levels between those patients with recurrence of atrial tachyarrhythmias and those without at 12 months | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- National Research Center for Preventive Medicine, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Davtyan K, Topchyan A, Brutyan H, Kalemberg E, Simonyan G, Serdyuk S, Kharlap M, Bazaeva E. Does cryoballoon ablation affect the symptom severity of atrial fibrillation? Insights from 12-months continuous cardiac monitoring. BMC Cardiovasc Disord. 2025 Sep 26;25(1):674. doi: 10.1186/s12872-025-05134-4. PMID 41013270